CLINICAL TRIAL: NCT02194764
Title: A Breath-based Naltrexone Adherence Tool to Manage Narcotic-addicted HIV Patients.
Brief Title: An Adherence Tool to Manage Narcotic -Addicted HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xhale Assurance (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: 2012115600086371; 1R43DA028740-01A1 (NIH)
Record Dates: First submitted 2014-07-15; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Naltrexone; 2-butanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Expirimental Formulation (Experimental): Participants will be administered a single encapsulated dose of the test formulation (Model Naltrexone 50mg containing 2-butanol). Breath samples will be taken over 90 minutes (-5, 0, 5, 10, 20, 40, 60, 90). Subjects will then be randomly crossed over to the four interventions (Formulation 1, Formulation 2, Formulation 3, Formulation-free positive control) three formulations from the first part of the study and a control administration (a capsule-in-capsule design).
  Interventions: Drug: Naltrexone and 2-butanol; Drug: 2-butanol which is encapsulated (size 3 capsule) plus 50 mg of naltrexone (HCl form)

INTERVENTIONS:
Drug: Naltrexone and 2-butanol — 50mg of Naltrexone and 40 or 80 mg of 2-butanol (depending on Stability Formulation in the first part of the study)
Drug: 2-butanol which is encapsulated (size 3 capsule) plus 50 mg of naltrexone (HCl form) — a capsule-in-capsule (CIC) design, will be prepared in the pharmacy by incorporating 40 or 80 mg (determined from the first part of the study) of 2-butanol which is encapsulated (size 3 capsule) plus 50 mg of naltrexone (HCl form) in a size 0 double blind hard gel capsule.

SUMMARY:
The purpose of this study is to develop a cost-effective breath-based medication adherence monitoring system that can monitor whether recovering opiate addicts actually take a specific treatment medication called naltrexone.

DETAILED DESCRIPTION:
This study will have two parts. In the first part we will create eight SMART capsule-based naltrexone systems using 4 general types of pharma formulation strategies. Model naltrexone (50mg) formulations containing the GRAS taggant, 2-butanol (40 or 80 mg) will be prepared and preliminary stability studies executed. Type 1 is a hydrophobic system, Type 2 is a hydrophilic system, Type 3 is a reverse micelle system and Type 4 is a water-in-oil microemulsion system. All formulations will be prepared using USP-grade excipients, 2-butanol, naltrexone base and naltrexone HCl. Naltrexone HCl has significant water solubility and will be used in the preparation of formulation types 2 and 4, whereas the more lipid soluble free base of naltrexone will be used in formulation types 1 and 3. Manufacturer's specifications supplied by Capsugel will be used to determine compatibility between the capsule material and the proposed excipients, and will guide capsule selection (gelatin or HPMC).Prepared formulations will be characterized by particle size analysis and analyzed to determine the actual concentrations of naltrexone and 2-butanol. Particle sizing will be accomplished by dynamic light scattering using a 90Plus particle size analyzer. With formulation types 1 and 2, the technique will demonstrate the homogeneity of the mixture and the absence of particulates. With types 3 and 4, particle size distributions will be measured to confirm the presence of monodisperse reverse micelles or nanoscale droplets. The concentration of naltrexone in each final formulation will be verified by Liquid chromatography-mass spectrometry (LC-MS) and /or Ultra Performance Liquid Chromatography (UPLC). The concentration of 2-butanol will be determined by gas chromatography-Mass Spectrometry (GC-MS). Following the initial characterization, the formulations will be stored in sealed vials and placed in ICH standard stability conditions and tested at weekly intervals over 1, 3 and 6 months. The three outstanding formulation candidates will be selected to use in part two of the study.

In the second part the three formulations will be selected from those meeting the criteria for stability, solubility, particle size, color and concentration of 2-butanol in the first part of the study. Each of these formulations will be prepared by a certified pharmacy. In addition to the three selected naltrexone formulations, a fourth dosage form, a capsule-in-capsule (CIC) design, will be prepared in the pharmacy by incorporating 40 or 80 mg (determined from the first part of the study) of 2-butanol which is encapsulated (size 3 capsule) plus 50 mg of naltrexone (HCI form) in a size 0 double blind hard gel capsule. This capsule-in-capsule design will serve as a formulation-free positive control.

Note: All naltrexone formulations, which will be administered to human subjects, will contain quantities of excipients/components already designated by the FDA as being safe (e.g., inactive ingredient list, permissible daily exposure [PDE], GRAS/direct food additive designation).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide written informed consent
* Subject is at least 18 Years of Age
* Subject must be willing to comply with study procedures

Exclusion Criteria:

* <18 years
* Subject has a history of opioid use disorder
* current chronic opioid therapy or recent (past week) acute opioid therapy,
* currently pregnant
* contraindications to naltrexone use per FDA label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Concentration of 2-butanol determined by gas chromatography mass spectroscopy (GC-MS) | Weekly intervals over 1, 3 and 6 months.
  The primary outcome is to identify three outstanding candidates based on physiochemical principles and the concentration of 2-butanol determined by GC-MS. Following the initial characterization, the formulations will be stored in sealed vials and placed in ICH standard stability conditions and tested at weekly intervals over 1, 3 and 6 months.
breath concentration versus time | -5, 0, 5, 10, 20, 40, 60, 90 min
  The relationship between the breath concentration (measured via mGC-MOS and gas chromatography mass spectroscopy [GC-MS]) of 2-butanol (taggant) and 2-butanone (metabolite) versus time will be determined after the oral administration of 3 promising naltrexone formulations selected from part of 1 of the study and a positive control.

SECONDARY OUTCOMES:
Breath Pharmacokinetics (Cmax) of the Naltrexone Formulations | -5, 0, 5, 10, 20, 40, 60, 90
  The secondary outcome will be to examine the breath pharmacokinetics of 2-butanol, 2-butanone, and cyclopropylcarboxaldehyde [CPCA, a natural metabolite of naltrexone] in human subjects following oral administration of the three selected naltrexone formulations or a positive control containing 2-butanol. Using an endpoint of differing CMAX in a repeated measures design, a difference in means of approximately 150 ppb (parts-per-million based on molar concentration [not mass]), a standard deviation of 75 ppb (based on pilot studies of oral capsules), 8 subjects per group are required (n=8/group) for a ANOVA repeated measures design with maximal tolerated Type I and II errors of 0.05 and 0.20.

CONTACTS AND LOCATIONS:
Overall Officials: Donn Dennis, M.D., F.A.H.A., Study Director — Xhale Smart, Inc.
Locations (1):
- University of Florida, Gainesville, Florida, United States